CLINICAL TRIAL: NCT03308045
Title: A Phase I/II, Open-label, Multicentre, Dose Escalation Study Assessing Safety/Tolerability of pEYS606 When Administered by Electrotransfer (ET) in Ciliary Muscle of Patients With Non-infectious Posterior, Intermediate or Panuveitis
Brief Title: Evaluation of EYS606 in Patients With Non-infectious Posterior, Intermediate or Panuveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eyevensys (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EYS606-CT1
Record Dates: First submitted 2017-03-31; First posted 2017-10-12 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Non-infectious Uveitis
Keywords: plasmid; electrotransfer; ciliary muscle; uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Intervention Model Description: Clinical trial with a single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pEYS606 (Experimental): Cohort 1 (pEYS606 lower dose); Cohort 2 (pEYS606 intermediate dose); Cohort 3 (pEYS606 higher dose); Extension Cohort (pEYS606 maximum tolerated dose)
  Interventions: Biological: pEYS606

INTERVENTIONS:
Biological: pEYS606 — pEYS606 is a DNA plasmid solution administered by electrotransfection into the ciliary muscle

SUMMARY:
Primary objective: safety and tolerability

Secondary objectives: additional indicators of long term safety and indicators of clinical activity

Exploratory objectives: to characterize EYS606 biodistribution, immunogenicity and biomarkers

DETAILED DESCRIPTION:
The maximum study duration per patient is 51 Weeks (including an up to 3 week screening period + 48 weeks follow-up after treatment).

The study is conducted in 2 parts. Part 1 is a dose escalation phase which will investigate three pEYS606 doses levels (lower, intermediate and higher dose) over 3 cohorts. Part 1 of the study has been completed. Part 2, the extension phase, which is now ongoing will confirm to safety of the maximum tolerated higher dose from Part 1 and allow a preliminary assessment of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 18 years of age or older
* Both female patients of childbearing potential and male patients able to father a child must agree to practice at least one effective method of birth control for six months following administration of study medication. Acceptable methods of birth control for this study include hormonal contraception (birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide or surgical sterilization (hysterectomy, tubal ligation or vasectomy). Patients with a hysterectomy or vasectomy (or have a partner with a hysterectomy or vasectomy) are exempt from using these methods of birth control.
* Female patients of childbearing potential must not be pregnant or breast-feeding and must have a negative urine pregnancy test at baseline and throughout the study.
* Voluntary written informed consent before performance of any study related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
* Patient has only one eligible eye with the following criteria:
* non-infectious intermediate, posterior, or panuveitis,
* media clarity, pupillary dilation, and individual cooperation sufficient for adequate fundus imaging,
* macular atrophy, AND/OR degenerative macular edema, AND/OR advanced optic neuropathy, AND/OR macular scar,
* Patients must maintain regiment of local and/or systemic corticosteroids between screening and baseline (if applicable).

Visual Criteria - Part 1 (enrolment is Part 1 is completed)

- BCVA of 0.1 (ETDRS of 35) or worse at screening in the treated eye, and BCVA of 0.32 or higher in the fellow eye.

Key Inclusion Criteria - Part 2 (enrolment in Part 2 is ongoing)

* BCVA of ≤ 0.63 or 20/32 Snellen but ≥ 0.025 or 20/800 Snellen (equivalent to ≥ 5 and ≤ 77 ETDRS letters) in the treated eye
* Patient must have a diagnosis of non-infectious uveitis of any anatomic subtype
* Patient must have a history of chronic or recurrent uveitis requiring or having required treatment with corticosteroids (systemic, periocular or intraocular) and/or systemic immunosuppressive medication(s) in the 12 months prior to the screening visit
* At the screening and baseline visits patient must have active uveitis as evidenced by at least one or more of the following in the study eye:

oActive retinal vasculitis (retinal vascular leakage) oVitreous haze grade ≥ 2+ oAnterior chamber cell grade ≥ 2+ oMacular edema

* Patient receiving concomitant topical and/or systemic corticosteroids or allowed systemic immunosuppressive medications must have maintained the same treatment regimen (dosage/frequency) for at least 2 weeks prior to the baseline (V1) visit, (if applicable).
* Willingness to receive local therapy to treat ocular inflammation in the fellow eye during the course of the study (if needed).

Exclusion Criteria:

* Patient has or is suspected to have infectious uveitis or a uveitis masquerade syndrome.
* Patient suspected to have tuberculosis, has had a positive test for tuberculosis in the past or has a positive γ-interferon tuberculosis test at the screening visit.
* For a patient with a primary diagnosis of idiopathic intermediate uveitis exclusion of any signs of multiple sclerosis must be demonstrated by an MRI examination of the brain and orbits with gadolinium prior to the baseline visit.
* Patient with macular edema as the only evidence of uveitis (e.g. absence of any vitreous haze or vasculitis) for which a non-uveitic cause of macular edema such as cataract extraction, age-related macular degeneration, diabetic retinopathy or retinal vein occlusion cannot be excluded.
* Patient with media opacity in the study eye that precludes visualization of the fundus or that is likely to require cataract surgery during the course of the trial.
* Patient with history of glaucoma filtering surgery (e.g. trabeculectomy or aqueous shunt implant) or who underwent eye surgery within 3 months in the treated eye.
* Patient who has uncontrolled intraocular pressure of ≥ 25 mmHg in the study eye at the screening and baseline visits.
* Patient with intraocular hypotension (<6 mmHg) that in the opinion of the Investigator would interfere with the administration of EYS606 or the evaluation of its safety or efficacy.
* Patient with history of scleritis, scleral thinning, cicatrizing conjunctival diseases, severe ocular allergies or other severe ocular surface disease that could interfere with the administration of EYS606 or the evaluation of its safety or efficacy.
* Patient has received Ozurdex® (dexamethasone implant) or other intraocular or periocular corticosteroids injections within 3 months prior to the baseline visit in the study eye
* Patient has received a fluocinolone implant (Retisert®, Illuvien®, YutiqTM) within 12 months prior to the baseline visit in the study eye.
* Patient has received treatment with a TNFα inhibitor intravitreally in the study eye within 2 months prior to the baseline visit.
* Patient has received intravitreal anti-VEGF therapy such as Lucentis® (ranibizumab) or Avastin® (bevacizumab) or Eylea® (aflibercept) within 2 months prior to the baseline visit or Beovu® (Brolucizumab) within 3 months prior to the baseline visit in the study eye.
* Patient has received intravitreal methotrexate within 2 months prior to the baseline visit in the study eye.
* Patient with a history of allergic reaction or intolerance to any routinely used ophthalmic medicines (e.g. fluorescein dye, topical dilating agents or local anesthetics) that will be prescribed during the course of the study.
* Patient with active or uncontrolled underlying systemic autoimmune or inflammatory disease requiring or likely to require an increase in systemic immunosuppressive medications or treatment with a biologic agent during the course of the study.
* Patient has received treatment with an alkylating agent (cyclophosphamide or chlorambucil) for the management of uveitis or an associated underlying disease.
* Patient has received treatment with a systemic biologic therapy (e.g. anti-TNFα, anti-IL-1, anti-IL-6, anti-IL-17, interferon) within 1 month prior to the baseline visit.
* Patient has received treatment with Rituximab within 6 months of the baseline visit.
* Patient with a history of or current evidence of any unstable medical condition (such as heart disease due to a cardiac conduction abnormality requiring a pacemaker, neurologic or psychiatric disorders requiring electroconvulsive therapy, acute or chronic liver diseases, malignancy, severe systemic allergy, etc.) that in the opinion of the Investigator, would expose the subject to an undue risk of a significant adverse event or interfere with the administration of EYS606 or the evaluation of its safety or efficacy during the course of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Number of patients with treatment emergent adverse events | 4 weeks
  Assessment of the safety and tolerability of EYS606

SECONDARY OUTCOMES:
Change from baseline in ocular safety assessments | 6 months
  Measured as change from baseline in adverse events, concomitant medications, intraocular pressure, electroretinogram, electrocardiogram, vital signs, physical exam and routine labs (blood and urinalysis)
Improvement in best corrected visual acuity | 6 months
  Measured as change from baseline eye in best corrected visual acuity using ETDRS scale
Improvement in anterior chamber cell grade | 6 months
  Measured as change from baseline in anterior cell grade according to the SUN scale
Improvement in vitreous haze grade | 6 months
  Measures as change from baseline in vitreous haze grade according to SUN scale
Improvement in central retinal thickness | 6 months
  Measures as change from baseline in central retinal thickness using ocular coherence tomography
Change in corticosteroid dose | 6 months
  Measures as change from baseline in prescribed dose of corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Antoine AB BREZIN, MD, Principal Investigator — Hôpital Cochin - Paris - France
Locations (4):
- France (2):
  - CHU de Grenoble - Hôpital Michallon, Grenoble
  - Hôpital Cochin, Paris
- United Kingdom (2):
  - Bristol Eye Hospital, Bristol
  - Moorfields Eye Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Touchard E, Benard R, Bigot K, Laffitte JD, Buggage R, Bordet T, Behar-Cohen F. Non-viral ocular gene therapy, pEYS606, for the treatment of non-infectious uveitis: Preclinical evaluation of the medicinal product. J Control Release. 2018 Sep 10;285:244-251. doi: 10.1016/j.jconrel.2018.07.013. Epub 2018 Aug 1. PMID 30009894